CLINICAL TRIAL: NCT05665153
Title: Symphony IL-6 Study in Patients at Risk of Severe Sepsis Due to COVID-19 and/or Influenza Infection
Brief Title: Symphony IL-6 Study in Patients at Risk of Severe Sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bluejay Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CES-0006_r2.1
Record Dates: First submitted 2022-12-07; First posted 2022-12-27 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Severe Sepsis
Keywords: SIRS; ARDS; COVID-19; Influenza A; Influenza Type B; Respiratory Failure
MeSH Terms: conditions — Sepsis; COVID-19; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Symphony IL-6 is a device that quantitates human IL-6 by fluorescence enzyme immunoassay (FEIA) from whole-blood specimens. Use of Symphony IL- 6 removes the need for plasma separation before testing. Symphony IL-6 comprises two components, the Symphony Fluorescence Immunoanalyzer and the Symphony IL-6 Cartridge. Whole blood is added to the cartridge and then up to six cartridges can be inserted into the immunoanalyzer. After 20 minutes a readout and printout are given with a quantitative IL-6 concentration. The used cartridges are fully enclosed and can be easily disposed of in general hospital bio-waste. Given the nature of this device and its portability, there is potential for future deployment in a near patient setting.

This study is to establish an interleukin-6 (IL-6) cutoff value using the Symphony IL-6 test for patients at high risk of severe sepsis caused by a COVID-19 and/or influenza infection.

ELIGIBILITY:
Inclusion Criteria:

* Whole-blood specimen collected in EDTA anticoagulant tube
* Subject is 22+ years of age
* A minimum volume of 0.3 ml blood will be collected for Symphony IL-6 testing
* Subjects who have concurrently received CRP test results
* Subject is confirmed to be COVID-19 positive by an EUA or FDA cleared SARS-CoV-2 positive RT-PCR test, and/or the subject is confirmed to be influenza-A or influenza-B positive by an FDA cleared test.

Exclusion Criteria:

* Subject is receiving an anti-IL-6 treatment
* Hemolyzed specimens

Min Age: 22 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: We will enroll approximately 200 individuals, whole-blood specimens collected as baseline samples from hospitalized individuals with confirmed COVID-19 and/or influenza patients at the University of Michigan Medical Center, Ann Arbor, MI.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-11-22 (Actual); Primary Completion 2024-08-21 (Estimated); Study Completion 2024-11-21 (Estimated)

PRIMARY OUTCOMES:
Concentration of IL-6 in hospitalized patients with COVID-19 and/or Influenza who require invasive mechanical ventilation | Total duration of COVID-19 and/or influenza hospitalization, up to 1 year
  Patients hospitalized with confirmed COVID-19 and/or influenza who require invasive mechanical ventilation due to complications with the infection.

SECONDARY OUTCOMES:
Concentration of IL-6 in hospitalized patients with COVID-19 and/or Influenza who expire during hospital stay | Total duration of COVID-19 and/or influenza hospitalization, up to 1 year
  Patients hospitalized with confirmed COVID-19 and/or influenza who expire during hospital stay.
Concentration of IL-6 in hospitalized patients with COVID-19 and/or Influenza who develop severe or critical illness | Total duration of the COVID-19 hospitalization, up to 1 year
  Severe Illness (any one of the following):
  1. SpO2 < 94% on room air at sea level
  2. Ratio of arterial partial pressure of oxygen to fraction of inspired oxygen (PaO2/FiO2) < 300 mmHg
  3. Respiratory frequency > 30 breaths/min
  4. Or lung infiltrates >50%
  Critical Illness (any one of the following):
  1. Respiratory failure
  2. Septic shock
  3. Multiple organ dysfunction

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan Medical Center, Ann Arbor, Michigan, United States